CLINICAL TRIAL: NCT00485095
Title: A Single Centre, Randomized Crossover Double-Blind Placebo-Controlled Study to Measure the Effect of Plant Sterol Supplement on Blood Cholesterol
Brief Title: The Effect of Plant Sterol Supplement on Blood Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Mills DA (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2.2006.3407
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2009-02

CONDITIONS: High Blood Cholesterol Level
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Behavioral: Intake of plant sterols

SUMMARY:
The purpose of this study is to determine whether supplement of plant sterol could lower blood cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-80 years old
* Total cholesterol: 4.5-7.5 mmol/l
* Triglycerides at or below 4.0 mmol/l

Exclusion Criteria:

* BMI at or above 35 kg/m2
* Secondary hyperlipidemia, included diabetes
* Hypertension (at og higher than 170/110)
* Coronar, perifery or cerebral vascular disease last 3 months
* Familial hypercholesterolemia
* Change in dose of statins, oestrogen or contraceptives last 3 months
* Taking drugs which are known to interfere with the plasma level of cholesterol
* Chronic rheumatoid diseases or other diseases known to affect c-reactive protein
* Pregnancy
* Lactation
* Planning to reduce weight
* Taking plant sterols

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Ose, MD, Principal Investigator — Lipidklinikken, Rikshospitalet-Radiumhospitalet HF
Locations (2):
- Norway (2):
  - Lipidklinikken, Rikshospitalet Radiumhospitalet HF, Oslo
  - Rikshospitalet Radiumhospitalet HF, Oslo, Norway, Oslo

REFERENCES:
- [Derived] Ottestad I, Ose L, Wennersberg MH, Granlund L, Kirkhus B, Retterstol K. Phytosterol capsules and serum cholesterol in hypercholesterolemia: a randomized controlled trial. Atherosclerosis. 2013 Jun;228(2):421-5. doi: 10.1016/j.atherosclerosis.2013.03.001. Epub 2013 Mar 20. PMID 23623012